CLINICAL TRIAL: NCT04988945
Title: Sequential TransArterial Chemoembolization and Stereotactic RadioTherapy Followed by Durvalumab (MEDI4736) and Tremelimumab for Downstaging Hepatocellular Carcinoma for Hepatectomy
Brief Title: TACE and SBRT Followed by Double Immunotherapy for Downstaging Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-046
Record Dates: First submitted 2021-06-29; First posted 2021-08-04 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: HCC
Keywords: HCC; TACE; SBRT; immunotherapy; hepatocellular carcinoma; liver cancer; unresectable; large liver tumour
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Tremelimumab (Experimental): 1500mg Durvalumab administered IV over 60 minutes on Day 1 of each immunotherapy treatment every 4 weeks until disease progression (PD) and 300mg Tremelimumab administered over 60 minutes on Day 1 of cycle 1.
  Interventions: Procedure: TACE; Radiation: SBRT; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Procedure: TACE — Procedure of TACE will be standardized.
Radiation: SBRT — SBRT screening and planning will be performed by radiation therapists, medical physicists, and oncologists.
Drug: Durvalumab — 1500mg Durvalumab administered IV over 60 minutes on Day 1 of each immunotherapy treatment every 4 weeks until disease progression (PD)
Drug: Tremelimumab — 300mg Tremelimumab administered over 60 minutes on Day 1 of cycle 1.

SUMMARY:
This study is a prospective phase II, single arm mono-institutional study conducted in Queen Mary Hospital (Hong Kong) assessing the efficacy and safety of the sequential administration of trans-arterial chemo-embolization (TACE) and stereotactic body radiotherapy (SBRT) with immune checkpoint inhibitors in unresectable hepatocellular carcinoma (HCC) patients.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a serious global health problem. It ranks the fifth in incidence and third in cancer-related mortality at Hong Kong in 2015. The disease has high mortality rate, and surgery is the only curative therapy although only 30% of patients are diagnosed early enough to undergo liver resection or transplantation or radiofrequency ablation (RFA). For inoperable patients with disease limited to liver, trans-arterial chemo-embolization (TACE) is the most commonly used therapy. Previous randomized studies have demonstrated its survival benefit, however it rarely cures the disease; also its efficacy is very limited in patients with sizable tumor or multi-focal diseases. Efforts have been made to improve the response of treatment, but none has consistently demonstrated the benefit. As a result, over the past decade, there is no major advancement in the treatment strategy for intermediate stage HCC patients. Recently, stereotactic body radiotherapy (SBRT) has emerged as one of the promising local therapy of HCC. This advanced radiotherapy technique allows killing of cancer cells by delivering a potent dose of radiation with excellent geometric precision. Data have demonstrated its favorable local control rate and toxicity profile in locally advanced HCC. Further, recent studies, including our series, indicated that combining SBRT and TACE is therapeutically superior. As such, it is postulated that combined TACE+SBRT is a more potent local therapy than TACE in preventing tumor progression, and it may potentially translate into survival benefit.

The recent discovery in immune-oncology represents another breakthrough in management of HCC. Pre-clinical data showed that there is high expression of immunosuppressive cells and up-regulation of programmed death receptor 1 (PD-1) and cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) immune checkpoints in the HCC microenvironment; it provides the rationale for immunotherapy to be used in this setting. This premise was supported by several early phase clinical studies, in which anti-PD-1/programmed death ligand 1 (PD-L1) therapy resulted in a durable response and favorable survival. More intriguingly, there are scientific and clinical data in supporting the synergy between immune checkpoint inhibitors (ICI) and SBRT for both local tumor regression and distant control (out-of-the-field abscopal) effect. For high risk HCC, such approach may warrant further exploration.

Based on all these, a hypothesis is made that combined TACE+SBRT followed by immunotherapy is a promising strategy in treating unresectable HCC. In this single-arm prospective phase II study, it is aimed at evaluating the efficacy and safety of this treatment regime.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Diagnosis of unresectable HCC confirmed pathologically or made according to

   American Association for the Study of Liver Diseases (AASLD) practice guideline 2010:

   patients with cirrhosis of any etiology and patients with chronic hepatitis B (HBV) who may not have fully developed cirrhosis, the presence of liver nodule >1cm and demonstrated in a single contrast-enhanced dynamic imaging [either computed tomography (CT) or magnetic resonance imaging (MRI)] of intense arterial uptake and "washout" in portal venous and delayed phases.
3. Adult male or female aged >18 years at time of study entry
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
5. Body weight >30kg
6. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
7. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
8. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
9. Must have a life expectancy of at least 12 weeks
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. Tumor size 5-25cm and number of lesions ≤3
12. Portal vein involvement (Vp1-3) is allowed: Vp1, presence of a tumor thrombus distal to, but not within, the second-order branches of the portal vein; Vp2, presence of a tumor thrombus in the second-order branches of the portal vein; Vp3, presence of a tumor thrombus in the first-order branches of the portal vein.
13. Liver volume minus gross tumor volume (GTV) > 700cc
14. Child-Pugh liver function class A-B7
15. No prior immunotherapy
16. Subjects with confirmed concomitant HBV infection (defined as HBsAg positive or HBV DNA detectable) that are eligible for inclusion must be treated with antiviral therapy (per local institutional practice) prior to enrollment to ensure adequate viral suppression (HBV DNA < 2000 IU/mL), must remain on antiviral therapy for the study duration, and continue therapy for 6 months after the last dose of investigational product(s)
17. At least one measurable lesion according to RECIST v1.1.

Adequate normal organ and marrow function as defined below:

* Haemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count (ANC ≥1.5 (or 1.0) x (> 1500 per mm^3)
* Platelet count ≥ 75 x 109/L (>75,000 per mm^3)
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
* AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
* Measured creatinine clearance (CL) >45 mL/min or Calculated creatinine clearance CL>45 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Participation in another clinical study with an investigational product within 4 weeks prior to the first dose of study treatment
2. Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study
3. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with Durvalumab or Tremelimumab may be included only after consultation with the Study Physician.
4. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.

   Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Prior radiotherapy to the region of liver or selective internal radiotherapy
6. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
7. History of primary immunodeficiency or allogenic organ transplantation.
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
10. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
11. History of leptomeningeal carcinomatosis
12. Presence of extra-hepatic metastases (M1). Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
13. Has untreated central nervous system (CNS) metastases and/or carcinomatous meningitis identified either on the baseline brain imaging (RECIST)) for details on the imaging modality) obtained during the screening period or identified prior to signing the ICF.
14. History of active primary immunodeficiency
15. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of Durvalumab or Tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note:

    Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of Durvalumab monotherapy or180 days after the last dose of Durvalumab + Tremelimumab combination therapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomisation or treatment in a previous Durvalumab and/or Tremelimumab clinical study regardless of treatment arm assignment.
21. Patients who have received prior anti-PD-1, anti-PD-L1 or anti-CTLA-4:

    * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    * Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
22. Contraindicated of SBRT:

    * Any one hepatocellular carcinoma > 25 cm
    * Total maximal sum of hepatocellular carcinoma > 30 cm
    * More than 3 discrete hepatic nodule
    * Direct tumor extension into the stomach, duodenum, small bowel, large bowel, common or main branch of biliary tree
23. Main portal vein, contralateral portal vein, (Vp4) or inferior vena cava (IVC) thrombosis / involvement
24. Presence of clinically meaningful ascites as ascites requiring non pharmacologic intervention (eg, paracentesis) or escalation in pharmacologic intervention to maintain symptomatic control
25. Hepatic encephalopathy
26. Active or prior documented gastrointestinal variceal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Downstaging for hepatectomy | From the date of first study treatment to the date of last study treatment, an average of 3 years
  To assess the number of patients amendable to curative surgical interventions (resection or radiofrequency ablation) after successful down-sizing of tumor(s) by intervention in HCC patients treated with combined TACE and SBRT followed by Durvalumab plus Tremelimumab

SECONDARY OUTCOMES:
Response rate measured by mRECIST criteria | From the date of screening to radiographically documented progression according to mRECIST 1.1, assessed up to 3 years
  Complete response (CR): Disappearance of any intra-tumoral arterial enhancement in all target lesions Partial response (PR): At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions Stable disease (SD): Any cases that do not qualify for either partial response or progressive disease Progressive disease (PD): An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started
Time to progression (TTP) | From the date of first study treatment to radiographically documented progression according to mRECIST 1.1, assessed up to 3 years
  measured from the date of first study treatment to radiographically documented progression according to mRECIST 1.1. This does not include death from any cause.
Progression-free survival (PFS) | From the date of first study treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause, whichever occurs first, assessed up to 3 years
  measured from the date of first study treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.
Overall survival (OS) | From the date of first study treatment to the date of death from any cause, assessed up to 5 years
  measured from date of first study treatment to the date of death from any cause
Toxicity tolerability measurement in treatment related procedure | From the date of screening to 90 days after last treatment, around 3 years and 90 days
  To measure the toxicities in HCC patients treated with combined TACE and SBRT followed by Durvalumab plus Tremelimumab. Dosage used will be recorded each time together with the response of patients. If any adverse event happens, the highest dosage will be noted down.
Questionnaire based Quality of Life (QoL) assessment | From the date of screening to radiographically documented progression according to mRECIST 1.1, an average of 3 years
  To evaluate the patient-reported quality of life (QoL) treated with combined TACE and SBRT followed by Durvalumab plus Tremelimumab. Questionnaires EORTC-QLQ-C30 and FACT Hep will be used
Pathological response | From the date of first study treatment to amendable to surgery after receiving combined TACE and SBRT followed by Durvalumab plus Tremelimumab, whichever occurs first, assessed up to 5 years
  Defined as the percentage of surface with non-viable cancer cells (represented by necrosis or fibrosis, the ultimate stage of necrosis) in relation to the total tumor area and will be equal to: 100% - viable cancer cells (%). If there are multiple tumors, the mean percentage will be used. Pathological complete response (pCR) is defined by the absence of viable tumor cells in any nodule.

CONTACTS AND LOCATIONS:
Overall Officials: Albert CHAN, Principal Investigator — Department of Surgery, The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Surgery, The University of Hong Kong, Hong Kong
  - The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawkins MA, Dawson LA. Radiation therapy for hepatocellular carcinoma: from palliation to cure. Cancer. 2006 Apr 15;106(8):1653-63. doi: 10.1002/cncr.21811. PMID 16541431
- [Background] Seong J, Kim SH, Suh CO. Enhancement of tumor radioresponse by combined chemotherapy in murine hepatocarcinoma. J Gastroenterol Hepatol. 2001 Aug;16(8):883-9. doi: 10.1046/j.1440-1746.2001.02533.x. PMID 11555102
- [Background] Chiang CL, Chan MKH, Yeung CSY, Ho CHM, Lee FAS, Lee VWY, Wong FCS, Blanck O. Combined stereotactic body radiotherapy and trans-arterial chemoembolization as initial treatment in BCLC stage B-C hepatocellular carcinoma. Strahlenther Onkol. 2019 Mar;195(3):254-264. doi: 10.1007/s00066-018-1391-2. Epub 2018 Nov 9. PMID 30413833
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Fife BT, Bluestone JA. Control of peripheral T-cell tolerance and autoimmunity via the CTLA-4 and PD-1 pathways. Immunol Rev. 2008 Aug;224:166-82. doi: 10.1111/j.1600-065X.2008.00662.x. PMID 18759926
- [Background] Stewart R, Morrow M, Hammond SA, Mulgrew K, Marcus D, Poon E, Watkins A, Mullins S, Chodorge M, Andrews J, Bannister D, Dick E, Crawford N, Parmentier J, Alimzhanov M, Babcook JS, Foltz IN, Buchanan A, Bedian V, Wilkinson RW, McCourt M. Identification and Characterization of MEDI4736, an Antagonistic Anti-PD-L1 Monoclonal Antibody. Cancer Immunol Res. 2015 Sep;3(9):1052-62. doi: 10.1158/2326-6066.CIR-14-0191. Epub 2015 May 5. PMID 25943534
- [Background] Tarhini AA, Kirkwood JM. Tremelimumab (CP-675,206): a fully human anticytotoxic T lymphocyte-associated antigen 4 monoclonal antibody for treatment of patients with advanced cancers. Expert Opin Biol Ther. 2008 Oct;8(10):1583-93. doi: 10.1517/14712598.8.10.1583. PMID 18774925
- [Background] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867